CLINICAL TRIAL: NCT01134185
Title: Evaluation of Pharmacokinetics, Safety and Tolerability of a Single Dose of Prucalopride, in Subjects With Moderate and Severe Hepatic Impairment, in Comparison With Healthy Subjects
Brief Title: Evaluation of Prucalopride in Subjects With Moderate and Severe Hepatic Impairment
Acronym: HI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M0001-C103
Record Dates: First submitted 2010-05-21; First posted 2010-05-31 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2011-10

CONDITIONS: Hepatic Impairment
Keywords: Two groups of 8 hepatically impaired subjects, one group of 8 matched healthy subjects
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Active Comparator): Moderate hepatic impairment (grade B)
  Interventions: Drug: prucalopride
- Group II (Active Comparator): Severe hepatic impairment (grade C)
  Interventions: Drug: prucalopride
- Group III (Active Comparator): healthy subjects
  Interventions: Drug: prucalopride

INTERVENTIONS:
Drug: prucalopride — single oral dose of 2 mg prucalopride
  Arms: Group I
Drug: prucalopride — single oral dose of 2 mg prucalopride
  Arms: Group II
Drug: prucalopride — single dose of 2 mg prucalopride
  Arms: Group III

SUMMARY:
This is a single centre, open-label phase I trial to investigate the effects of moderate to severe hepatic impairment on the pharmacokinetics of prucalopride in comparison with healthy volunteers. Furthermore the short-term safety and tolerability of a single dose of prucalopride will be assessed.

DETAILED DESCRIPTION:
In this phase I trial two groups of 6 to 8 hepatically impaired subjects will be evaluated. The first group are the moderate hepatic impairment (Grade B) subjects and the second group the severe hepatic impairment (grade C) subjects. Subjects for both groups will be recruited and treated in parallel. After all subjects with hepatic impairment completed the treatment a third group with matching healthy volunteers will be recruited. Eight healthy subjects will be selected matching for age, gender and weight (BMI based).

The subjects will receive a single dose of 2 mg prucalopride in the morning after overnight fasting followed by the consumption of a standard breakfast after 2 hours.

Pharmacokinetic evaluation of blood samples will be done immediately before and at a specific timepoint up to 120h post-dosing. Urine samples will be taken to determine prucalopride.

Adverse events, including serious adverse events, will be reported from signing the Informed Consent until the last visit. Safety blood samples and a urine sample for urinalysis will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Main inclusion criteria for hepatic impairment subjects:

  * Moderate (Grade B) or severe (Grade C) chronic hepatic impairment according to Child-Pugh classification; Hepatic impairment must be stable, both clinically and biochemically;
  * Within the normal range of body height and weight on the basis of the Body Mass Index.
* Main inclusion criteria for healthy subjects:

  * Matching on sex, age and weight(BMI based).

Exclusion Criteria:

* History or suspicion of barbiturate, amphetamine or narcotic abuse; Suspicion of current alcohol abuse;
* Clinical suspicion or laboratory evidence of unstable hepatic impairment or acute liver injury;
* Clinically relevant renal disease as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 6 days
  Evaluation of prucalopride in blood immediately before and at 17 timepoints post dosing and in urine at 8 collection time points.

SECONDARY OUTCOMES:
Safety and tolerability | 6 days
  Evaluation of safety parameters by measuring adverse events, safety, blood and urine samples, ECGs, vital signs and physical examinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow, Russia